CLINICAL TRIAL: NCT06866704
Title: Pulsed-Field Ablation Vs. Radiofrequency Ablation CombIned with Vein of Marshall Ethanol Ablation on Mitral Isthmus Block and Clinical Outcomes in Persistent Atrial Fibrillation: the PRIME-AF Randomized Clinical Trial
Brief Title: Pulsed-Field Ablation Vs. Radiofrequency Ablation CombIned with Vein of Marshall Ethanol Ablation on Mitral Isthmus Block and Clinical Outcomes in Persistent Atrial Fibrillation
Acronym: PRIME-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: lingzhiyu (Other)
Responsible Party: Sponsor-Investigator, lingzhiyu, Director, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIME-AF
Record Dates: First submitted 2025-03-01; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF)
Keywords: persistent atrial fibrillation; pulsed field ablation; EI-VOM
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pulsed field ablation (Experimental): patients receive pulsed field ablation (PFA) to achieve pulmonary vein isolation (PVI), circumferential BOX ablation around bilateral pulmonary veins, and mitral isthmus ablation.
  Interventions: Procedure: catheter ablation
- EI-VOM (Placebo Comparator): anhydrous alcohol is first injected into the Marshall vein, followed by radiofrequency catheter ablation to complete PVI, BOX lesion sets, and mitral isthmus ablation.
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — In the experimental group, patients receive pulsed field ablation (PFA) to achieve pulmonary vein isolation (PVI), circumferential BOX ablation around bilateral pulmonary veins, and mitral isthmus ablation. In the control group, anhydrous alcohol is first injected into the Marshall vein, followed by radiofrequency catheter ablation to complete PVI, BOX lesion sets, and mitral isthmus ablation.

SUMMARY:
Atrial fibrillation (AF) is one of the most common clinical arrhythmias, and catheter ablation serves as a critical therapeutic approach. For persistent atrial fibrillation, several proposed ablation strategies-including the 2C3L technique, BOX lesion sets, and substrate modification-remain highly controversial regarding long-term success rates. Multiple studies suggest that linear ablation beyond pulmonary vein isolation (PVI) often fails to achieve durable block due to incomplete ablation lines, which significantly contributes to postoperative recurrence of atrial arrhythmias.

In recent years, electrophysiologists have explored various methods to improve mitral isthmus (MI) ablation, such as combined endo-epicardial ablation and radiofrequency ablation (RFA) combined with Marshall vein alcohol ablation. While RFA combined with anhydrous alcohol injection into the Marshall vein enhances MI block rates, it is associated with prolonged procedure time, unpredictable ablation zones, and higher complication risks (e.g., coronary artery spasm, pericarditis).

Pulsed field ablation (PFA), an emerging non-thermal ablation technology, offers potential advantages such as tissue selectivity, shorter procedure time, and fewer complications. Studies report that RFA achieves near 100% immediate block rates; however, there is a lack of sufficient comparative studies on the efficacy and safety between these two ablation approaches. This study aims to compare the clinical outcomes and safety profiles of PFA versus RFA combined with Marshall vein alcohol injection in patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent atrial fibrillation;
2. Ejection fraction >30%;
3. NYHA functional class I-III;
4. Left atrial diameter <55 mm on echocardiography;
5. Signed informed consent form;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with a life expectancy of less than 2 years due to non-cardiovascular factors;
3. Uncontrolled hyperthyroidism, severe liver or kidney dysfunction;
4. History of atrial fibrillation ablation;
5. History of heart transplantation, complex congenital heart disease, or rheumatic heart disease;
6. Contraindications to contrast agents, radiofrequency ablation, antiarrhythmic drugs, or anticoagulants;
7. Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular 8.accident within 12 weeks prior to enrollment;

9.Other conditions deemed unsuitable for participation by investigators; 10.Participation in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate success rate of mitral isthmus ablation block | immediately after the procedure
  Bidirectional MI block was confirmed by the following criteria: (1) proximal-to-distal CS activation pattern when pacing at the left lateral ridge; (2) longer SA interval at the left lateral ridge when pacing at the distal CS compared to pacing at the proximal CS
Mitral isthmus block rate | 20 minutes after the procedure
  Bidirectional MI block was confirmed by the following criteria: (1) proximal-to-distal CS activation pattern when pacing at the left lateral ridge; (2) longer SA interval at the left lateral ridge when pacing at the distal CS compared to pacing at the proximal CS

SECONDARY OUTCOMES:
The incidence of atrial arrhythmias (tachycardia, atrial flutter, atrial fibrillation) over 30 seconds without antiarrhythmic drugs was followed up for 12 months. | 1 year
  The incidence of atrial arrhythmias (tachycardia, atrial flutter, atrial fibrillation) over 30 seconds without antiarrhythmic drugs was followed up for 12 months.
time of operation | immediately after the procedure
  Total operating time,Ablation time,Mitral isthmus ablation time,Radiation time;
complication | 2 weeks after the procedure
  Incidence of pericardial tamponade, acute heart failure, pericardial effusion, pleural effusion; Puncture complications; Incidence of cerebral infarction and TIA; Death;

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davong B, Adelino R, Delasnerie H, Albenque JP, Combes N, Cardin C, Voglimacci-Stephanopoli Q, Combes S, Boveda S. Pulsed-Field Ablation on Mitral Isthmus in Persistent Atrial Fibrillation: Preliminary Data on Efficacy and Safety. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 2):1070-1081. doi: 10.1016/j.jacep.2023.03.021. Epub 2023 Jun 21. PMID 37354173
- [Background] Sang C, Liu Q, Lai Y, Xia S, Jiang R, Li S, Guo Q, Li Q, Gao M, Guo X, Huang L, Liu N, Jiang C, Zuo S, Liu X, Li M, Ge W, Song S, Chen L, Xie S, Zou J, Chen K, Liu X, Hu H, Wang X, Zhang J, Wang Z, Wang C, He L, Jiang C, Tang R, Zhou N, Wang Y, Long D, Du X, Jiang C, Macle L, Dong J, Ma C; PROMPT-AF investigators. Pulmonary Vein Isolation With Optimized Linear Ablation vs Pulmonary Vein Isolation Alone for Persistent AF: The PROMPT-AF Randomized Clinical Trial. JAMA. 2025 Feb 4;333(5):381-389. doi: 10.1001/jama.2024.24438. PMID 39556379
- [Background] Valderrabano M, Peterson LE, Swarup V, Schurmann PA, Makkar A, Doshi RN, DeLurgio D, Athill CA, Ellenbogen KA, Natale A, Koneru J, Dave AS, Giorgberidze I, Afshar H, Guthrie ML, Bunge R, Morillo CA, Kleiman NS. Effect of Catheter Ablation With Vein of Marshall Ethanol Infusion vs Catheter Ablation Alone on Persistent Atrial Fibrillation: The VENUS Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1620-1628. doi: 10.1001/jama.2020.16195. PMID 33107945